CLINICAL TRIAL: NCT01857310
Title: Folic Acid and Zinc Supplementation Trial: A Multi-center, Double-blind, Block-randomized, Placebo-controlled Trial
Brief Title: Folic Acid and Zinc Supplementation Trial (FAZST)
Acronym: FAZST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAZST
Record Dates: First submitted 2013-05-13; First posted 2013-05-20 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Pregnancy; Live Birth; Spontaneous Abortion
Keywords: Folic Acid; Zinc; Semen; In vitro fertilization; Assisted reproductive technology; Ovulation induction; Intrauterine insemination; Pregnancy; Live Birth; Abortion, spontaneous
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Folic acid and zinc supplementation (Experimental): 5 mg folic acid and 30 mg elemental zinc, taken orally, daily for 6 months.
  Interventions: Dietary Supplement: 5 mg folic acid and 30 mg elemental zinc
- Placebo (Placebo Comparator): Matching placebo, taken orally daily for 6 months.
  Interventions: Drug: Placebo Comparator: Placebo

INTERVENTIONS:
Dietary Supplement: 5 mg folic acid and 30 mg elemental zinc
  Arms: Folic acid and zinc supplementation
Drug: Placebo Comparator: Placebo
  Arms: Placebo

SUMMARY:
The overarching goal of this trial is to determine if an intervention comprising folic acid and zinc dietary supplementation improves semen quality and indirectly fertility outcomes (i.e., live birth rate) among couples trying to conceive and seeking assisted reproduction. The following study objectives underlie successful attainment of the overarching research goal:

1. To estimate the effect of folic acid and zinc dietary supplementation on semen quality parameters, including but not limited to concentration, motility, morphology, and sperm DNA integrity, relative to the placebo group.
2. To estimate the effect of folic acid and zinc dietary supplementation on fertility treatment outcomes [fertilization, embryo quality, implantation/human Chorionic Gonadotropin (hCG) confirmed pregnancy, clinical pregnancy, live birth], relative to the placebo group.
3. To estimate the association between semen quality parameters, sperm DNA integrity and fertility treatment outcomes (fertilization, embryo quality, clinical pregnancy, live birth) and to identify the best combination of semen quality parameters for prediction of clinical pregnancy and live birth.
4. To estimate the effect of folic acid and zinc dietary supplementation on fertilization rates among couples undergoing assisted reproductive technology procedures, relative to the placebo group.
5. To estimate the effect of folic acid and zinc dietary supplementation on embryonic quality among couples undergoing assisted reproductive technology procedures, relative to the placebo group.

DETAILED DESCRIPTION:
Two micronutrients fundamental to the process of spermatogenesis, folic acid (folate) and zinc, are of particular interest for fertility as they are of low cost and wide availability. Though the evidence has been inconsistent, small randomized trials and observational studies show that folate and zinc have biologically plausible effects on spermatogenesis and improved semen parameters. These results support the potential benefits of folate on spermatogenesis and suggest that dietary supplementation with folate and zinc may help maintain and improve semen quality, and perhaps, fertility rates.

The Epidemiology Branch of the Eunice Kennedy Shriver National Institute of Child Health and Human Development intends to conduct a multi-site double-blind, randomized controlled clinical trial to evaluate the effect of folic acid and zinc dietary supplementation on semen quality and conception rates among male partners of couples seeking assisted reproduction. Randomization will be stratified (with random sequences of block sizes) by site and assisted reproduction technique (IVF, non-IVF receiving fertility treatment at a study site, and non-IVF receiving fertility treatment at a nonstudy site) to ensure that balance between the treatment groups is maintained within site and within fertility treatment type over the enrollment period.

The study is designed with a sample size of 2,400 randomized participants based on obtaining adequate power to detect meaningful differences in the live birth rate between cohorts. Since the comparison of sperm parameters are differences between continuous assay measurements, this sample size will be more than sufficient for the primary sperm parameter comparisons. Additionally, calculations were done to demonstrate adequate statistical power when stratified analysis is to be performed (i.e., sample size distributions among the strata and their corresponding live birth RRs detected at 80% statistical power, with an alpha level of 0.05 and a total sample size of 2400 couples divided among the folic acid/zinc and placebo arms of the trial).

Data collection will include screening male and female partners for eligibility, administering baseline questionnaires, and collecting biospecimens in both partners of the couple, body measurements for both partners, daily journal reporting for male partners, medical record abstraction related to required treatment and outcome data, and semen quality of four samples collected at baseline, two, four, and six months following study enrollment. A data coordinating center (DCC) will support the trial.

The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two cohorts based on the randomized assignment, both overall and by treatment strata (IVF, non-IVF receiving fertility treatment at a study site, and non-IVF receiving fertility treatment at a nonstudy site).This approach will be applied to the two primary endpoints (semen parameters and live birth rate) as well as designated secondary endpoints (number of follicles, number and proportion of oocytes fertilized).

The DCC will perform periodic safety analyses and present interim reports to the Data and Safety Monitoring Board (DSMB) as requested, during the recruitment phases of the trial. It is anticipated that safety analyses will be performed every 6-12 months. The final analysis will be performed upon completion of data collection and editing in the follow-up and close-out phase of the trial. Also one full formal interim analysis is planned and the power calculations with considerations for the choice of optimal time for the analysis have been conducted.

ELIGIBILITY:
Couples Inclusion Criteria:

1. Heterosexual couples in a committed relationship with a female partner aged 18-45 years and male partner aged 18 years and older attempting to conceive and seeking assisted reproduction at participating fertility clinics.
2. Couples actively trying to conceive.
3. Couples who are planning ovulation induction (OI), natural fertility optimization methods, or intrauterine insemination (IUI) should be willing to be on the study dietary supplement for at least 3 weeks before starting the next assisted reproduction cycle.Women with regular periods may initiate their fertility therapy at the start of the woman's menstrual cycle following randomization if randomization occurred within the first 10 days of the cycle, but must wait one menstrual cycle if the visit occurred after day 10 of the cycle). For women with irregular periods or amenorrhea, the male must be on the study supplement for 3 weeks prior to initiation of any ovulation induction medication (e.g., clomid, letrozole, gonadotropins).

Couples Exclusion Criteria:

1. Female partner unwilling to participate (e.g., no abstraction of her assisted fertility treatment record or unwilling to complete baseline visit).
2. Couples using donor, cryopreserved sperm, or sperm obtained via microsurgical or percutaneous epididymal sperm aspiration.
3. Couples attempting to conceive with a gestational carrier (surrogate).
4. Positive urine pregnancy test at screening.

Male Inclusion Criteria:

1. Willing to provide semen samples according to the proposed schedule at baseline, 2, 4, and 6 months of follow-up.
2. Able to complete regular study questionnaires and daily journals aimed at capturing ejaculation, sexual intercourse and lifestyle factors considered to affect male fecundity (e.g., cigarette smoking, fever, high temperature environment and other environmental exposures) and other data collection instruments (e.g., physical activity, food frequency questionnaire, stress).

Male Exclusion Criteria:

1. Age <18 years.
2. Unwilling to abstain from use of non-study approved dietary supplements or medications containing folic acid or oral preparations containing zinc throughout the study.
3. Unwilling to abstain from use of testosterone supplementation throughout the study.
4. Diagnosis of Vitamin B12 deficiency or pernicious anemia.
5. Consuming a vegan diet.
6. A known genetic cause of male factor subfertility, including chromosomal disorders related to subfertility (e.g., Y chromosome deletions).
7. Males currently using and unwilling (or unable) to discontinue the following drugs known to interact with folic acid or interfere with the biosynthesis of folic acid will be excluded.

   1. Dihydrofolate reductase inhibitors: Trimethoprim, Triamterene, Bactrim, Iclaprim
   2. Sulfonamides: Hydrochlorothiazide (HCTZ), Metolazone, Indapamide, Lasix, Bumex, Torsemide, Chlorthalidone, Acetazolamide, Mefruside, Xipamide
   3. Sulfonylureas: Glipizide, Glyburide
   4. Cox-2 inhibitors: Celecoxib
   5. Others: Valproic acid, Probenecid, Sulfasalazine, Sumatriptan, Mafenide, Ethoxzolamide, Sulfiram, Zonisamide, Dorzolamide (optic), Dichlorphenamide, Fluorouracil, Capecitabine, Methotrexate
8. History of organ transplantation.
9. Physician diagnosed:

   1. Current poorly controlled chronic diseases such as heart disease, diabetes mellitus, hypertension, cancer, inflammatory diseases, autoimmune, thyroid disease, endocrine dysfunction, liver disease, kidney disease, or HIV/AIDS or other immune-insufficient related illnesses.
   2. Crohn's disease, celiac disease, ulcerative colitis, gastric bypass surgery, lap band surgery or history of intestinal surgery to remove a portion of small bowel. History of diseases/symptoms that require folic acid dietary supplementation, such as megaloblastic anemia, homocystinemia, and homocystinuria.
   3. History of alcohol dependency disorder and/or other drug/substance dependency in the past 180 days.
   4. History of psychoses or other mental conditions that would result in cognitive impairment and inability to participate in any part of this study including the informed consent process, as diagnosed by a physician within the past year.
10. History of vasectomy without reversal, obstructive azoospermia such as Congenital Bilateral Aplasia of Vas Deferens (CBAVD), or ejaculatory duct obstruction.
11. Known allergy to folic acid or zinc dietary supplements.

Female Exclusion Criteria:

Age <18 or >45 years.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2370 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique F. Schisterman, PhD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Sunni L. Mumford, PhD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); C. Matthew Peterson, MD, Principal Investigator — University of Utah; Jared C. Robins, MD, Principal Investigator — Northwestern University; Ginny L. Ryan, MD, MA, Principal Investigator — University of Iowa; Bradley J. Van Voorhis, MD, Principal Investigator — University of Iowa
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Center for Reproductive Medicine, Minneapolis, Minnesota
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] DiTosto JD, Caniglia EC, Hinkle SN, Sealy N, Schisterman EF, Johnstone E, Mendola P, Mills J, Hotaling J, Ryan G, Mumford SL. Target trial emulation of preconception serum vitamin D status on fertility outcomes: a couples-based approach. Fertil Steril. 2025 Feb;123(2):300-312. doi: 10.1016/j.fertnstert.2024.08.332. Epub 2024 Aug 20. PMID 39173703
- [Derived] DeVilbiss EA, Sjaarda LA, Peterson CM, Hotaling JM, Mills JL, Mendola P, Carrell DT, Johnstone E, Chen Z, Perkins NJ, Ryan G, Schisterman EF, Mumford SL. Longitudinal semen parameter assessments and live birth: variability and implications for treatment strategies. Fertil Steril. 2022 Nov;118(5):852-863. doi: 10.1016/j.fertnstert.2022.08.012. Epub 2022 Oct 1. PMID 36192231
- [Derived] Jenkins T, Aston K, Carrell D, DeVilbiss E, Sjaarda L, Perkins N, Mills JL, Chen Z, Sparks A, Clemons T, Chaney K, Peterson CM, Emery B, Hotaling J, Johnstone E, Schisterman E, Mumford SL. The impact of zinc and folic acid supplementation on sperm DNA methylation: results from the folic acid and zinc supplementation randomized clinical trial (FAZST). Fertil Steril. 2022 Jan;117(1):75-85. doi: 10.1016/j.fertnstert.2021.09.009. Epub 2021 Oct 14. PMID 34656303
- [Derived] Schisterman EF, Sjaarda LA, Clemons T, Carrell DT, Perkins NJ, Johnstone E, Lamb D, Chaney K, Van Voorhis BJ, Ryan G, Summers K, Hotaling J, Robins J, Mills JL, Mendola P, Chen Z, DeVilbiss EA, Peterson CM, Mumford SL. Effect of Folic Acid and Zinc Supplementation in Men on Semen Quality and Live Birth Among Couples Undergoing Infertility Treatment: A Randomized Clinical Trial. JAMA. 2020 Jan 7;323(1):35-48. doi: 10.1001/jama.2019.18714. PMID 31910279
- See also: The FAZST trial home page — https://www.nichd.nih.gov/about/org/diphr/officebranch/eb/folic-acid-zinc

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only the male partners in couples attempting to conceive were enrolled and assigned to treatment arms.
Groups:
- Folic Acid and Zinc Supplementation: 5 mg folic acid and 30 mg elemental zinc, taken orally, daily for 6 months.
  5 mg folic acid and 30 mg elemental zinc
- Placebo: Matching placebo, taken orally daily for 6 months.
  Placebo Comparator: Placebo
Period: Primary Analysis: Live Birth
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Started | 1185 (Male partner) | 1185 (Male partner)
Completed | 1185 (Chart abstraction of whether live birth occurred) | 1185 (Chart abstraction of whether live birth occurred)
Not Completed | 0 | 0
Period: Secondary Analysis: Semen Quality at 6m
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Started | 1185 (Male partner) | 1185 (Male partner)
Completed | 870 (Completed 6-month study visit) | 903 (Completed 6-month study visit)
Not Completed | 315 | 282
Not completed — Lost to Follow-up | 315 | 282

BASELINE CHARACTERISTICS:
Population: Only male partners randomized to each folic acid/zinc (n = 1185) and placebo (n = 1185) arms
Units Other Than Participants: Male-female couples
Groups:
- Total: Total of all reporting groups
Arm/Group | Folic Acid and Zinc Supplementation | Placebo | Total
Number analyzed (Participants) | 2370 | 2370 | 4740
Number analyzed (Male-female couples) | 1185 | 1185 | 2370
Age, Continuous [Mean (Standard Deviation); unit: years] — Male partner age, continuous Population: Male partners
  years
    number analyzed (Participants) | 1185 | 1185 | 2370
    (all) | 32.5 (5.7) | 32.7 (6.0) | 32.6 (5.9)
Age, Continuous [Mean (Standard Deviation); unit: years] — Female partner age, continuous Population: Female partners
  years
    number analyzed (Participants) | 1185 | 1185 | 2370
    (all) | 30.6 (5.0) | 30.8 (5.2) | 30.7 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1185 | 1185 | 2370
  Male | 1185 | 1185 | 2370
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Male partner race/ethnicity, customized Population: Male partners
  Participants
    number analyzed (Participants) | 1185 | 1185 | 2370
    Non-Hispanic white | 974 | 962 | 1936
    Non-Hispanic black | 21 | 34 | 55
    Asian | 43 | 46 | 89
    Hispanic or Latino | 70 | 68 | 138
    Other racial/ethnic groups | 74 | 68 | 142
    Do not wish to provide | 3 | 7 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Female partner race/ethnicity, customized Population: Female partners
  Participants
    number analyzed (Participants) | 1185 | 1185 | 2370
    Non-Hispanic white | 994 | 962 | 1956
    Non-Hispanic black | 22 | 21 | 43
    Asian | 61 | 70 | 131
    Hispanic or Latino | 52 | 75 | 127
    Other racial/ethnic groups | 51 | 50 | 101
    Do not wish to provide | 5 | 7 | 12
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Male partner body mass index Population: Male partners
  kg/m^2
    number analyzed (Participants) | 1185 | 1185 | 2370
    (all) | 30.1 (6.7) | 29.6 (6.7) | 29.8 (6.7)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Male partner systolic blood pressure Population: Male partners
  mmHg
    number analyzed (Participants) | 1185 | 1185 | 2370
    (all) | 126.8 (12.8) | 126.5 (13.9) | 126.7 (13.4)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Male partner diastolic blood pressure Population: Male partners
  mmHg
    number analyzed (Participants) | 1185 | 1185 | 2370
    (all) | 78.4 (10.8) | 78.0 (10.9) | 78.2 (10.9)
Education [Count of Participants; unit: Participants] — Male partner education Population: Male partners
  Participants
    number analyzed (Participants) | 1185 | 1185 | 2370
    High school or less | 198 | 173 | 371
    Some college | 428 | 386 | 814
    Bachelor's degree | 335 | 389 | 724
    Master's degree or higher | 212 | 220 | 432
    Do not wish to provide | 12 | 17 | 29
Employment status [Count of Participants; unit: Participants] — Male partner employment status Population: Male partners: 89 participants in the FA/Zn arm and 90 participants in the placebo arm did not provide this information.
  Participants
    number analyzed (Participants) | 1096 | 1095 | 2191
    Not employed | 149 | 148 | 297
    Employed part-time | 58 | 53 | 111
    Employed full-time | 802 | 798 | 1600
    Full-time student | 87 | 96 | 183
Marital status [Count of Units; unit: Male-female couples] — Population: Measure assessed among each of 2370 male-female couples (n=1185 active and 1185 placebo)
  Male-female couples
    number analyzed (Participants) | 1185 | 1185 | 2370
    Married/living with partner | 1180 | 1179 | 2359
    Single/other | 4 | 4 | 8
    Do not wish to provide | 1 | 2 | 3
Annual household income [Count of Units; unit: Male-female couples] — Population: Measure assessed among each of 2370 male-female couples (n=1185 active and 1185 placebo)
  Male-female couples
    number analyzed (Participants) | 1185 | 1185 | 2370
    <$40,000 | 176 | 157 | 333
    $40,000-$74,999 | 422 | 456 | 878
    $75,000-$99,999 | 261 | 232 | 493
    $100,000 and greater | 252 | 278 | 530
    Do not wish to provide | 74 | 62 | 136
Taking multivitamin within past 3 mo [Count of Participants; unit: Participants] — Male partner taking multivitamin within past 3 mo Population: Male partners: 434 participants in the FA/Zn arm and 433 participants in the placebo arm did not provide this information.
  Participants
    number analyzed (Participants) | 751 | 752 | 1503
    Yes | 298 | 284 | 582
    No | 453 | 468 | 921
Male factor infertility diagnosis [Count of Participants; unit: Participants] — Baseline male factor infertility diagnosis includes low sperm count, low sperm motility, abnormal morphology, poor DNA fragmentation, testicular failure, and other. Population: Male partners: 427 participants in the FA/Zn arm and 426 participants in the placebo arm did not provide this information.
  Participants
    number analyzed (Participants) | 758 | 759 | 1517
    No | 598 | 594 | 1192
    Yes | 160 | 165 | 325
Male health insurance [Count of Participants; unit: Participants] — Population: Male partners: 12 participants in the FA/Zn arm and 14 participants in the placebo arm did not provide this information.
  Participants
    number analyzed (Participants) | 1173 | 1171 | 2344
    Yes | 1108 | 1117 | 2225
    No | 65 | 54 | 119
Male infertility insurance [Count of Participants; unit: Participants] — Population: Male partners: 79 participants in the FA/Zn arm and 69 participants in the placebo arm did not provide this information.
  Participants
    number analyzed (Participants) | 1106 | 1116 | 2222
    Yes | 297 | 266 | 563
    No | 493 | 495 | 988
    Do not know | 316 | 355 | 671
Time trying to conceive [Median (Inter-Quartile Range); unit: months] — Population: Measure assessed among each of 2370 male-female couples (n=1185 active and 1185 placebo): 83 couples in the FA/Zn arm and 80 couples in the placebo arm did not provide this information.
  months
    number analyzed (Participants) | 1102 | 1105 | 2207
    number analyzed (Male-female couples) | 1102 | 1105 | 2207
    (all) | 19 [12 to 36] | 18 [12 to 36] | 18 [12 to 36]

OUTCOME MEASURES:

1. Primary Outcome: Live Birth
Description: Based on hospital delivery records
Time Frame: At delivery
Population: Complete randomized cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 1185 | 1185
Participants
  Overall | 404 | 416
  IVF stratum: number analyzed (Participants) | 185 | 188
  IVF stratum | 97 | 91
  Other treatment onsite: number analyzed (Participants) | 831 | 827
  Other treatment onsite | 264 | 277
  Other treatment offsite: number analyzed (Participants) | 169 | 170
  Other treatment offsite | 43 | 48
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Live birth will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Risk Difference (RD) = -0.9, 95% CI 2-sided [-4.7 to 2.8] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.88 to 1.09] — Adjusted for infertility treatment stratum and study site

2. Primary Outcome: Semen Volume
Description: Volume of the ejaculate, mL Assessed utilizing the World Health Organization (WHO) semen analysis procedure 5th edition World Health Organization. WHO laboratory manual for the Examination and processing of human semen. 5th Edition ed. Switzerland: 2010.
Time Frame: 6 months
Population: Analyzed overall and by fertility treatment stratum (subgroup) 870 and 903 men in the active and placebo treatment arms, respectively, returned for the 6-month study visit. 76 men in the active arm and 67 men in the placebo arm did not provide semen samples at this visit.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 794 | 836
mL
  Overall | 3.5 (1.7) | 3.5 (1.8)
  IVF stratum: number analyzed (Participants) | 124 | 135
  IVF stratum | 3.5 (1.5) | 3.5 (1.7)
  Other treatment onsite: number analyzed (Participants) | 566 | 590
  Other treatment onsite | 3.5 (1.7) | 3.5 (1.8)
  Other treatment offsite: number analyzed (Participants) | 104 | 110
  Other treatment offsite | 3.5 (1.7) | 3.4 (1.7)
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Semen volume will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.2 to 0.2] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.1 to 0.2] — Weighted for loss to follow-up and adjusted for infertility treatment stratum and study site

3. Primary Outcome: Sperm Concentration
Description: Number of spermatozoa per unit of volume of semen Assessed utilizing the World Health Organization (WHO) semen analysis procedure 5th edition World Health Organization. WHO laboratory manual for the Examination and processing of human semen. 5th Edition ed. Switzerland: 2010.
Time Frame: 6 months
Population: 870 and 903 men in the active and placebo treatment arms, respectively, returned for the 6-month study visit. 76 men in the active arm and 67 men in the placebo arm did not provide semen samples at this visit. Additionally, one male participant in the placebo arm had insufficient quantity or quality to assess concentration.
Measure: Mean (Standard Deviation); unit: 10^6 spermatozoa/mL
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 794 | 835
10^6 spermatozoa/mL
  Overall | 84.8 (85.2) | 89.0 (85.0)
  IVF stratum: number analyzed (Participants) | 124 | 135
  IVF stratum | 81.8 (96.5) | 76.1 (78.6)
  Other treatment onsite: number analyzed (Participants) | 566 | 590
  Other treatment onsite | 85.0 (83.1) | 92.2 (84.8)
  Other treatment offsite: number analyzed (Participants) | 104 | 110
  Other treatment offsite | 87.2 (83.0) | 87.7 (92.5)
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. The confidence interval for sperm concentration represents 95.1% coverage to properly account for the alpha spent in the interim analysis; Test type: Superiority; Mean Difference (Final Values) = -4.3, 95.1% CI 2-sided [-12.5 to 3.9] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -5.2, 95.1% CI 2-sided [-13.6 to 3.1] — Weighted for loss to follow-up and adjusted for fertility treatment stratum and study site

4. Primary Outcome: Sperm Motility
Description: % motile (including percentage of progressive motile sperm and percentage of nonprogressive motile sperm) Assessed utilizing the World Health Organization (WHO) semen analysis procedure 5th edition World Health Organization. WHO laboratory manual for the Examination and processing of human semen. 5th Edition ed. Switzerland: 2010.
Time Frame: 6 months
Population: 870 and 903 men in the active and placebo treatment arms, respectively, returned for the 6-month study visit. 76 men in the active arm and 67 men in the placebo arm did not provide semen samples at this visit. Additionally, one male participant in the placebo arm had insufficient quantity or quality to assess motility.
Measure: Mean (Standard Deviation); unit: % motile
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 794 | 835
% motile
  Overall | 52.7 (21.2) | 53.2 (20.1)
  IVF stratum: number analyzed (Participants) | 124 | 135
  IVF stratum | 51.7 (21.9) | 51.7 (20.0)
  Other treatment onsite: number analyzed (Participants) | 566 | 590
  Other treatment onsite | 52.5 (21.1) | 53.9 (19.5)
  Other treatment offsite: number analyzed (Participants) | 104 | 110
  Other treatment offsite | 55.0 (20.9) | 51.5 (22.8)
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. The confidence interval for sperm motility represents 95.1% coverage to properly account for the alpha spent in the interim analysis; Test type: Superiority; Mean Difference (Final Values) = -0.5, 95.1% CI 2-sided [-2.5 to 1.5] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -0.6, 95.1% CI 2-sided [-2.7 to 1.4] — Weighted for loss to follow-up and adjusted for infertility treatment stratum and study site

5. Primary Outcome: Sperm Morphology
Description: % normal morphology Assessed utilizing the World Health Organization (WHO) semen analysis procedure 5th edition World Health Organization. WHO laboratory manual for the Examination and processing of human semen. 5th Edition ed. Switzerland: 2010.
Time Frame: 6 months
Population: 870 and 903 men in the active and placebo treatment arms, respectively, returned for the 6-month study visit. 76 men in the active arm and 67 men in the placebo arm did not provide semen samples at this visit. Additionally, 19 men in the active arm and 17 men in the placebo arm had insufficient quantity or quality to assess morphology.
Measure: Mean (Standard Deviation); unit: % normal
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 775 | 819
% normal
  Overall | 5.7 (4.2) | 6.0 (4.8)
  IVF stratum: number analyzed (Participants) | 124 | 135
  IVF stratum | 5.2 (4.3) | 5.4 (4.7)
  Other treatment onsite: number analyzed (Participants) | 566 | 590
  Other treatment onsite | 5.6 (4.0) | 6.2 (4.9)
  Other treatment offsite: number analyzed (Participants) | 104 | 110
  Other treatment offsite | 6.7 (4.9) | 5.6 (4.3)
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. The confidence interval for sperm morphology represents 95.1% coverage to properly account for the alpha spent in the interim analysis; Test type: Superiority; Mean Difference (Final Values) = -0.4, 95.1% CI 2-sided [-0.8 to 0.1] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -0.4, 95.1% CI 2-sided [-0.9 to 0] — Weighted for loss to follow-up and adjusted for infertility treatment stratum and study site

6. Primary Outcome: DNA Fragmentation Index
Description: Comet assay used to measure sperm DNA integrity based on excess DNA strand breaks Assessed utilizing the World Health Organization (WHO) semen analysis procedure 5th edition World Health Organization. WHO laboratory manual for the Examination and processing of human semen. 5th Edition ed. Switzerland: 2010.
Time Frame: 6 months
Population: 870 and 903 men in the active and placebo treatment arms, respectively, returned for the 6-month study visit. 76 men in the active arm and 67 men in the placebo arm did not provide semen samples at this visit. Additionally, 44 men in the active arm and 55 men in the placebo arm had insufficient quantity or quality to assess DFI.
Measure: Mean (Standard Deviation); unit: % breakage
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 750 | 781
% breakage
  Overall | 29.7 (20.5) | 27.2 (17.8)
  IVF stratum: number analyzed (Participants) | 124 | 135
  IVF stratum | 27.1 (19.6) | 26.8 (19.6)
  Other treatment onsite: number analyzed (Participants) | 566 | 590
  Other treatment onsite | 30.0 (20.3) | 27.0 (16.8)
  Other treatment offsite: number analyzed (Participants) | 104 | 110
  Other treatment offsite | 30.7 (22.7) | 28.5 (20.5)
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. DNA fragmentation will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [0.5 to 4.4] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [0.3 to 4.3] — Weighted for loss to follow-up and adjusted for infertility treatment stratum and study site

7. Primary Outcome: Total Motile Sperm Count
Description: Calculated as semen volume (mL) * sperm concentration (10^6 spermatozoa/mL) * motility (% motile)
Time Frame: 6 months
Population: 870 and 903 men in the active and placebo treatment arms, respectively, returned for the 6-month study visit. 76 men in the active arm and 67 men in the placebo arm did not provide semen samples at this visit. Additionally, 1 man in the active arm and 2 men in the placebo arm had insufficient quantity or quality to assess total motile count.
Measure: Mean (Standard Deviation); unit: million motile sperm
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 793 | 834
million motile sperm
  Overall | 183 (226) | 182 (212)
  IVF stratum: number analyzed (Participants) | 124 | 135
  IVF stratum | 165 (221) | 152 (188)
  Other treatment onsite: number analyzed (Participants) | 566 | 590
  Other treatment onsite | 186 (226) | 188 (207)
  Other treatment offsite: number analyzed (Participants) | 104 | 110
  Other treatment offsite | 192 (233) | 184 (262)
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Total motile sperm count will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-19.7 to 22.5] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-20.9 to 21.4] — Weighted for loss to follow-up and adjusted for infertility treatment stratum and study site

8. Secondary Outcome: Human Chorionic Gonadotropin (hCG) Detected Pregnancy (Implantation)
Description: A quantitative hCG evaluation in serum > 5 milli-international units per milliliter (mIU/ml)
Time Frame: For IVF, 12 days post embryo transfer for day 5 embryo transfers, and 14 days post embryo transfer for day 3 embryo transfers; for couples undergoing OI/IUI, after self-report of positive pregnancy test
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 1185 | 1185
Participants | 479 | 490
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. hCG detected pregnancy will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Risk Difference (RD) = -0.9, 95% CI 2-sided [-4.7 to 3.0] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.91 to 1.09] — Adjusted for infertility treatment stratum and study site

9. Secondary Outcome: Clinical Intrauterine Pregnancy
Description: Visualized gestational sac in the uterus on ultrasound
Time Frame: approximately 6.5 weeks gestation
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 1185 | 1185
Participants | 449 | 462
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Clinical intrauterine pregnancy will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Risk Difference (RD) = -1.0, 95% CI 2-sided [-4.9 to 2.8] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.89 to 1.08] — Adjusted for infertility treatment stratum and study site

10. Secondary Outcome: Ectopic Pregnancy
Description: Either visualization of no gestational sac in the uterus with a suspicious mass in the adnexa on ultrasound, an hCG level more than 1500 mIU/ml without visualization of an intrauterine gestational sac on ultrasound, or a slowly rising or plateauing serum hCG level without visualization of an intrauterine gestation on ultrasound.
Time Frame: approximately 6.5 weeks gestation
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 1185 | 1185
Participants | 6 | 5
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Ectopic pregnancy will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Risk Difference (RD) = 0.1, 95% CI 2-sided [-0.5 to 0.6] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 1.21, 95% CI 2-sided [0.37 to 3.97] — Adjusted for fertility treatment stratum and study site

11. Secondary Outcome: Early Pregnancy Loss
Description: hCG pregnancy loss will be defined as a serum hCG > 5 mIU/ml followed by a decline. Clinically recognized pregnancy losses will be defined as visualization of an intrauterine gestational sac followed by a loss prior to 20 weeks gestation.
Time Frame: hcG-detected pregnancy until 20 weeks of pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 1185 | 1185
Participants | 137 | 150
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Early pregnancy loss will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Risk Difference (RD) = -1.1, 95% CI 2-sided [-3.7 to 1.5] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.75 to 1.15] — Adjusted for infertility treatment stratum and study site

12. Secondary Outcome: Preeclampsia or Gestational Hypertension
Description: Abstracted from hospital records and medical charts
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 1185 | 1185
Participants | 47 | 51
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Preeclampsia/gestational hypertension will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Risk Difference (RD) = -0.3, 95% CI 2-sided [-1.9 to 1.3] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.63 to 1.36] — Adjusted for infertility treatment stratum and study site

13. Secondary Outcome: Gestational Diabetes
Description: Abstracted from hospital records and medical charts
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 1185 | 1185
Participants | 26 | 34
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Gestational diabetes will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Risk Difference (RD) = -0.7, 95% CI 2-sided [-1.9 to 0.6] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.77, 95% CI 2-sided [0.47 to 1.27] — Adjusted for infertility treatment stratum and study site

14. Secondary Outcome: Cesarean Delivery
Description: Abstracted from hospital records and medical charts
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 1185 | 1185
Participants | 143 | 129
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Cesarean delivery will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Risk Difference (RD) = 1.2, 95% CI 2-sided [-1.4 to 3.8] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 1.12, 95% CI 2-sided [0.89 to 1.39] — Adjusted for infertility treatment stratum and study site

15. Secondary Outcome: Preterm Delivery
Description: Abstracted from hospital records and medical charts
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 1185 | 1185
Participants | 67 | 45
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Preterm delivery will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Risk Difference (RD) = 1.9, 95% CI 2-sided [0.2 to 3.6] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 1.49, 95% CI 2-sided [1.04 to 2.16] — Adjusted for infertility treatment stratum and study site

16. Secondary Outcome: Small for Gestational Age
Description: Abstracted from hospital records and medical charts
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 1185 | 1185
Participants | 62 | 59
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Small for gestational age will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Risk Difference (RD) = 0.3, 95% CI 2-sided [-1.5 to 2.0] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.75 to 1.49] — Adjusted for infertility treatment stratum and study site

17. Secondary Outcome: Gestational Age
Description: Abstracted from hospital records and medical charts
Time Frame: Delivery
Population: Among participants with live birth
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 404 | 416
weeks | 38.6 (2.5) | 38.8 (2.2)
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Gestational age will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Risk Difference (RD) = -0.2, 95% CI 2-sided [-0.5 to 0.1] — Adjusted for infertility treatment stratum and study site

18. Secondary Outcome: Birth Weight
Description: Abstracted from hospital records and medical charts
Time Frame: Delivery
Population: Among participants with live birth
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 404 | 416
grams | 3062 (731) | 3133 (654)
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Birth weight will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Risk Difference (RD) = -64.7, 95% CI 2-sided [-156 to 26.4] — Adjusted for infertility treatment stratum and study site

19. Secondary Outcome: Stillbirth
Description: Loss at or after 20 weeks gestation. Determined based on hospital records and medical chart abstraction.
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 1185 | 1185
Participants | 1 | 4
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Stillbirth will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Risk Difference (RD) = -0.2, 95% CI 2-sided [-0.6 to 0.1] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.25, 95% CI 2-sided [0.03 to 2.24] — Adjusted for infertility treatment stratum and study site

20. Secondary Outcome: Neonatal Mortality
Description: Abstracted from hospital records and medical charts
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 1185 | 1185
Participants | 3 | 2
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Neonatal mortality will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Risk Difference (RD) = 0.1, 95% CI 2-sided [-0.3 to 0.5] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 1.50, 95% CI 2-sided [0.25 to 8.95] — Adjusted for infertility treatment stratum and study site

21. Secondary Outcome: Major Neonatal Complications
Description: Abstracted from hospital records and medical charts: includes bronchopulmonary dysplasia, necrotizing enterocolitis, severe intraventricular hemorrhage, periventricular leukomalacia, and retinopathy of prematurity
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 1185 | 1185
Participants | 2 | 1
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Major neonatal complications will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Risk Difference (RD) = 0.1, 95% CI 2-sided [-0.2 to 0.4] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 1.99, 95% CI 2-sided [0.18 to 21.9] — Adjusted for infertility treatment stratum and study site

22. Secondary Outcome: Structural Malformations
Description: Abstracted from birth record: includes major (n = 21; 6 with known genetic cause), minor (n = 6), and unclassified (n = 2) defects Structural birth defects: includes hydronephrosis/ureteropelvic junction obstruction, transposition of the great arteries, renal agenesis, cleft lip, club feet, multicystic/dysplastic kidney, tetralogy of fallot, gastroschisis, atrioventricular septal defects, other oral-facial defects, other cardiovascular defects, other CNS defects, other eye defects, other oral-facial defects, other anomalies, other syndromes
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 1185 | 1185
Participants | 15 | 14
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Structural malformations will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Risk Difference (RD) = 0.1, 95% CI 2-sided [-0.8 to 1.0] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.53 to 2.21] — Adjusted for infertility treatment stratum and study site

23. Secondary Outcome: Severe Maternal Morbidity
Description: Abstracted from delivery record: including postpartum hemorrhage, anemia requiring transfusion, sepsis, seizure, HELLP syndrome or preeclampsia with pulmonary edema
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 1185 | 1185
Participants | 15 | 10
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Severe maternal morbidity will be compared using two sided tests conducted at the 0.05 level; Test type: Superiority; Risk Difference (RD) = 0.4, 95% CI 2-sided [-0.4 to 1.3] — Adjusted for infertility treatment stratum and study site
Statistical Analysis 2: Comparison: Folic Acid and Zinc Supplementation vs Placebo; [analysis description as in outcome 23, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 1.50, 95% CI 2-sided [0.68 to 3.32] — Adjusted for infertility treatment stratum and study site

24. Secondary Outcome: Fertilization Rate Per Cycle, %
Description: Among participants in the IVF stratum Oocytes will be assessed 16-18 hours after insemination or microinjection to determine whether fertilization occurred. Fertilization will be considered normal if two pronuclei and two polar bodies are identified. Oocytes without visible pronuclei will be considered unfertilized. Oocytes with more than two pronuclei will be considered abnormally fertilized, and will thus be discarded.
Time Frame: Up to 9 months of fertility treatment post-randomization
Population: 124 and 135 participants randomized to active and placebo arms, respectively Fertilization rate unavailable in medical records for 17 and 28 participants in the active and placebo arms, respectively
Measure: Mean (Standard Deviation); unit: percent per cycle
Units Other Than Participants: cycles
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 107 | 107
Number analyzed (cycles) | 124 | 119
percent per cycle | 75.3 (2.25) | 77.7 (1.74)
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Fertilization rate will be compared using generalized estimating equations accounting for multiple cycles per couple; Test type: Superiority; Mean Difference (Final Values) = -2.34, 95% CI 2-sided [-7.90 to 3.23]

25. Secondary Outcome: Number of Good Quality Embryos on Day 5 Per Cycle
Description: Among participants in the IVF stratum For couples who meet criteria for blastocyst culture, embryos will be graded 5 days after fertilization based on Society for Assisted Reproductive Technologies (SART) morphology criteria.
Time Frame: Up to 9 months of fertility treatment post-randomization
Population: 124 and 135 participants randomized to active and placebo arms, respectively Day 5 good quality embryos unavailable in medical records for 56 and 64 participants in the active and placebo arms, respectively
Measure: Mean (Standard Deviation); unit: embryos per cycle
Units Other Than Participants: cycles
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 68 | 71
Number analyzed (cycles) | 72 | 74
embryos per cycle | 2.66 (0.23) | 2.98 (0.21)
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Number of good quality embryos will be compared using Poisson regression with generalized estimating equations accounting for multiple cycles per couple; Test type: Superiority; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.33 to 0.11]

26. Secondary Outcome: Percentage of Good Quality Embryos on Day 5 Per Cycle
Description: as for outcome 25
Time Frame: Up to 9 months of fertility treatment post-randomization
Population: 124 and 135 participants randomized to active and placebo arms, respectively Proportion day 5 good quality embryos unavailable in medical records for 17 and 28 participants in the active and placebo arms, respectively
Measure: Mean (Standard Deviation); unit: percent per cycle
Units Other Than Participants: cycles
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 107 | 107
Number analyzed (cycles) | 124 | 119
percent per cycle | 17.2 (2.05) | 18.5 (1.81)
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Proportion of good quality embryos on day 5 will be compared using generalized estimating equations accounting for multiple cycles per couple; Test type: Superiority; Mean Difference (Final Values) = -1.31, 95% CI 2-sided [-6.66 to 4.05]

27. Secondary Outcome: Number of Embryos Transferred Per Cycle
Description: Among participants in the IVF stratum
Time Frame: Up to 9 months of fertility treatment post-randomization
Population: 124 and 135 participants randomized to active and placebo arms, respectively Proportion day 5 good quality embryos unavailable in medical records for 7 and 9 participants in the active and placebo arms, respectively
Measure: Mean (Standard Deviation); unit: embryos per cycle
Units Other Than Participants: cycles
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 117 | 126
Number analyzed (cycles) | 147 | 152
embryos per cycle | 1.50 (0.06) | 1.51 (0.05)
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Number of embryos transferred will be compared using Poisson regression with generalized estimating equations accounting for multiple cycles per couple; Test type: Superiority; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.11 to 0.10]

28. Secondary Outcome: Number of Embryos Cryopreserved Per Cycle
Description: Among participants in the IVF stratum
Time Frame: Up to 9 months of fertility treatment post-randomization
Population: 124 and 135 participants randomized to active and placebo arms, respectively Number of embryos cryopreserved unavailable in medical records for 40 and 35 participants in the active and placebo arms, respectively
Measure: Mean (Standard Deviation); unit: embryos per cycle
Units Other Than Participants: cycles
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 84 | 100
Number analyzed (cycles) | 92 | 116
embryos per cycle | 4.22 (0.32) | 4.32 (0.31)
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Number of embryos cryopreserved will be compared using Poisson regression with generalized estimating equations accounting for multiple cycles per couple; Test type: Superiority; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.23 to 0.18]

29. Secondary Outcome: Sperm Penetration Per Cycle, %
Description: Among participants in the IVF stratum
Time Frame: Up to 9 months of fertility treatment post-randomization
Population: 124 and 135 participants randomized to active and placebo arms, respectively Sperm penetration & unavailable in medical records for 114 and 121 participants in the active and placebo arms, respectively
Measure: Mean (Standard Deviation); unit: percent penetration
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 10 | 14
percent penetration | 62.7 (13.0) | 74.8 (11.0)
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Sperm penetration percentage will be compared using generalized estimating equations accounting for multiple cycles per couple; Test type: Superiority; Mean Difference (Final Values) = -12.1, 95% CI 2-sided [-45.4 to 21.2]

30. Secondary Outcome: Cells on Day 3 Per Embryo Per Cycle
Description: Among participants in the IVF stratum
Time Frame: Up to 9 months of fertility treatment post-randomization
Population: 1215 embryos among cycles among women in the FA/Zn arm; 1129 embryos among cycles among women in the placebo arm 124 and 135 participants randomized to active and placebo arms, respectively
  # of cells on day 3 unavailable in medical records for 25 and 36 participants in the active and placebo arms, respectively
Measure: Mean (Standard Deviation); unit: cells per embryo
Units Other Than Participants: cycles
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 99 | 99
Number analyzed (cycles) | 117 | 114
cells per embryo | 5.60 (0.20) | 5.98 (0.19)
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Number of cells on day 3 will be compared with Poisson regression using generalized estimating equations accounting for multiple embryos per cycle and multiple cycles per couple; Test type: Superiority; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.16 to 0.03]

31. Secondary Outcome: Cells on Day 3 Per Embryo Per Cycle, Categorical
Description: Number of cells per embryo among women in the IVF stratum
Time Frame: Up to 9 months of fertility treatment post-randomization
Population: 1222 embryos among cycles among women in the FA/Zn arm; 1140 embryos among cycles among women in the placebo arm 124 and 135 participants randomized to active and placebo arms, respectively
  # of cells on day 3 (categorical) unavailable in medical records for 25 and 36 participants in the active and placebo arms, respectively
Measure: Number; unit: predicted probability
Units Other Than Participants: cycles
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 99 | 99
Number analyzed (cycles) | 114 | 114
predicted probability
  Fewer than 4 cells | 0.27 | 0.22
  4 cells or greater | 0.73 | 0.78
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Number of cells on day 3 will be compared using generalized estimating equations accounting for multiple embryos per cycle and multiple cycles per couple; Test type: Superiority; Risk Ratio (RR) = 1.19, 95% CI 2-sided [0.88 to 1.61] — Fewer than 4 cells

32. Secondary Outcome: Cells on Day 5 Per Embryo Per Cycle, Categorical
Description: Among participants in the IVF stratum
Time Frame: Up to 9 months of fertility treatment post-randomization
Population: 1160 embryos among cycles among women in the FA/Zn arm and 1205 embryos among cycles among women in the placebo arm 124 and 135 participants randomized to active and placebo arms, respectively
  # of cells on day 5 (categorical) unavailable in medical records for 5 and 14 participants in the active and placebo arms, respectively
Measure: Number; unit: predicted probability
Units Other Than Participants: cycles
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 119 | 121
Number analyzed (cycles) | 141 | 141
predicted probability
  Fewer than 8 cells | 0.20 | 0.19
  8 cells or greater | 0.80 | 0.81
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Number of cells on day 5 will be compared using generalized estimating equations accounting for multiple embryos per cycle and multiple cycles per couple; Test type: Superiority; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.77 to 1.43] — Fewer than 8 cells

33. Secondary Outcome: Embryo Morphology on Day 3 Per Cycle, Categorical
Description: Among participants in the IVF stratum Embryos will be scored three days after fertilization according to the size and shape of blastomeres and to their degree of fragmentation.
  Veeck LL. Oocyte assessment and biological performance. Ann N Y Acad Sci 1988;541:259-74.:259-74.
Time Frame: Up to 9 months of fertility treatment post-randomization
Population: 961 embryos among cycles among women in the FA/Zn arm; 931 embryos among cycles among women in the placebo arm 124 and 135 participants randomized to active and placebo arms, respectively Embryo morphology on day 3 (categorical) unavailable in medical records for 27 and 37 participants in the active and placebo arms, respectively
Measure: Number; unit: predicted probability
Units Other Than Participants: cycles
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 97 | 98
Number analyzed (cycles) | 141 | 141
predicted probability
  Excellent or good | 0.66 | 0.68
  Fair or poor | 0.34 | 0.32
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Embryo morphology on day 3 will be compared using generalized estimating equations accounting for multiple embryos per cycle and multiple cycles per couple; Test type: Superiority; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.87 to 1.09] — Excellent or good morphology

34. Secondary Outcome: Embryo Morphology on Day 5 Per Cycle, Categorical
Description: as for outcome 25
Time Frame: Up to 9 months of fertility treatment post-randomization
Population: 973 embryos among cycles among women in the FA/Zn arm; 1009 embryos among cycles among women in the placebo arm 124 and 135 participants randomized to active and placebo arms, respectively Embryo morphology on day 5 (categorical) unavailable in medical records for 10 and 19 participants in the active and placebo arms, respectively
Measure: Number; unit: predicted probability
Units Other Than Participants: cycles
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 114 | 116
Number analyzed (cycles) | 132 | 134
predicted probability
  Excellent or good | 0.28 | 0.35
  Fair or poor | 0.72 | 0.65
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Embryo morphology on day 5 will be compared using generalized estimating equations accounting for multiple embryos per cycle and multiple cycles per couple; Test type: Superiority; Risk Ratio (RR) = 0.82, 95% CI 2-sided [0.63 to 1.06] — Excellent or good morphology

35. Secondary Outcome: Method of Fertilization Per Cycle
Description: Among participants in the in vitro fertilization (IVF) stratum: method of fertilization classified into intracytoplasmic sperm injection (ICSI) and other
Time Frame: Up to 9 months of fertility treatment post-randomization
Population: 1689 embryos among cycles among women in the active treatment arm; 1800 embryos among cycles among women in the placebo arm 124 and 135 participants randomized to active and placebo arms, respectively Method of fertilization unavailable in medical records for 2 and 5 participants in the active and placebo arms, respectively
Measure: Number; unit: predicted probability
Units Other Than Participants: cycles
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 122 | 130
Number analyzed (cycles) | 145 | 157
predicted probability
  ICSI | 0.74 | 0.79
  Other | 0.26 | 0.21
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Method of fertilization will be compared using generalized estimating equations accounting for multiple embryos per cycle and multiple cycles per couple; Test type: Superiority; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.80 to 1.09] — ICSI

36. Secondary Outcome: Quality of Embryos Transferred Per Cycle, Categorical
Description: Among participants in the IVF stratum Embryonic grading based on Society for Assisted Reproductive Technologies (SART) morphology criteria
Time Frame: Up to 9 months of fertility treatment post-randomization
Population: 172 embryos among cycles among women in the FA/Zn arm; 187 embryos among cycles among women in the placebo arm 124 and 135 participants randomized to active and placebo arms, respectively Quality of embryos transferred (categorical) unavailable in medical records for 21 and 30 participants in the active and placebo arms, respectively
Measure: Number; unit: predicted probability
Units Other Than Participants: cycles
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 103 | 105
Number analyzed (cycles) | 121 | 125
predicted probability
  Excellent or good | 0.75 | 0.73
  Fair or poor | 0.25 | 0.27
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Quality of embryos transferred will be compared using generalized estimating equations accounting for multiple embryos per cycle and multiple cycles per couple; Test type: Superiority; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.88 to 1.21] — Excellent or good quality

37. Secondary Outcome: Chromosomal Complement of Embryo Per Cycle
Description: Among participants in the IVF stratum Chromosomal complement in the embryo assessed using methodology cited by Rubio et al.
  Rubio C, Rodrigo L, Mir P et al. Use of array comparative genomic hybridization (array-CGH) for embryo assessment: clinical results. Fertil Steril 2013 March 15;99(4):1044-8.
Time Frame: Up to 9 months of fertility treatment post-randomization
Population: 124 and 135 participants randomized to active and placebo arms, respectively Chromosomal complement of embryo unavailable in medical records for 121 and 124 participants in the active and placebo arms, respectively
Measure: Number; unit: predicted probability
Units Other Than Participants: cycles
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
Number analyzed (Participants) | 3 | 11
Number analyzed (cycles) | 5 | 17
predicted probability
  Abnormal | 0.75 | 0.32
  Normal | 0.25 | 0.68
Statistical Analysis 1: Comparison: Folic Acid and Zinc Supplementation vs Placebo; The primary analysis plan is based on an "intention-to-treat" (ITT) approach comparing the two treatment arms based on the randomized assignment. The common null hypothesis states that the effect of folic acid/zinc on the outcomes is null compared to the placebo. Chromosomal complement will be compared using generalized estimating equations accounting for multiple cycles per couple; Test type: Superiority; Risk Ratio (RR) = 2.35, 95% CI 2-sided [0.74 to 7.43] — Abnormal

38. Other Pre Specified Outcome: Reproductive Hormones and Other Measured Biomarkers
Description: Urinary, serum, and salivary concentrations of reproductive hormones, particularly androgens, proteomic analysis of human sperm and cardiometabolic risk factors and markers of oxidative stress, as well as measures of trace elements in toenails (collected at month 4 clinic visit). Biospecimens have been collected but laboratory analysis still needs to be done to be able to evaluate these endpoints.
Time Frame: 4 or 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 6 month duration of the study.
Description: Adverse events were only collected from the male partners.
Arm/Group | Folic Acid and Zinc Supplementation | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1185 | 0/1185
Serious Adverse Events (participants affected / at risk) | 7/1185 | 5/1185
Other Adverse Events (participants affected / at risk) | 189/1185 | 162/1185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Folic Acid and Zinc Supplementation (N=1185) | Placebo (N=1185)
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hospitalisation (Surgical and medical procedures) | 1 | 0
Variococele repair (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Folic Acid and Zinc Supplementation (N=1185) | Placebo (N=1185)
Abdominal discomfort or pain (Gastrointestinal disorders) | 66 | 40
Pyrexia (General disorders) | 66 | 62
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 57 | 60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/10/NCT01857310/Prot_SAP_000.pdf